CLINICAL TRIAL: NCT02981953
Title: TRI-REPAIR: TrIcuspid Regurgitation RePAIr With CaRdioband Transcatheter System
Acronym: TRI-REPAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR1-1
Record Dates: First submitted 2016-11-20; First posted 2016-12-05 (Estimated); Results first posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Tricuspid Valve Insufficiency; Tricuspid Regurgitation; Tricuspid Valve Regurgitation; Cardiovascular Diseases; Heart Valve Diseases; Heart Diseases; Cardiac Valve Annuloplasty
Keywords: Valtech Cardio; Cardioband; Tricuspid
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Cardiovascular Diseases; Heart Valve Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardioband Tricuspid procedure (Other): Tricuspid valve repair with Cardioband implanted via transcatheter procedure under transesophageal echocardiography (TEE) and fluoroscopy guidance
  Interventions: Device: Cardioband Tricuspid

INTERVENTIONS:
Device: Cardioband Tricuspid — The Cardioband Adjustable implant is delivered and anchored to the tricuspid valve annulus by a transfemoral delivery system. The Cardioband TR will be deployed and adjusted under trans-esophageal and fluoroscopy guidance.

SUMMARY:
The current management of tricuspid regurgitation (TR) is either conservative (by medication) or by surgery, usually in concomitant with other valves repair or replacement. TR can worsen or appear late after successful mitral valve surgery which portends a poor prognosis. However, standard surgical approaches requiring cardiopulmonary bypass and especially second surgery have an excessive risks. Thus many patients are denied surgery because of unfavorable risk-benefit balance. Therefore there is a need for novel devices enabling interventional cardiologists and cardiothoracic surgeons to perform tricuspid annuloplasty by transcatheter methods. Cardioband replicates established surgical techniques (e.g., annuloplasty) using transfemoral approach, without sutures and with adjusted on the beating heart. Similar to the approved indication for mitral annuloplasty. The Cardioband System is expected to allow for treatment of patients that would otherwise not undergo Tricuspid valve repair due to the invasiveness of current techniques.

DETAILED DESCRIPTION:
The Cardioband Transcatheter System (Cardioband) is a marketed system that was approved for treatment of secondary (functional) mitral regurgitation (FMR) (CE granted on September 2015). The Cardioband is an annuloplasty band that is similar to a surgical annuloplasty, however deployed on the beating heart through a transvenous approach. The CE mark study with 30 subjects has been completed and documented significant reduction of severity of MR and improvement in quality of life by Minnesota living with heart failure questionnaire (MLHFQ), New York Heart Association (NYHA) and 6- minute walk test (6MWT), in subjects with moderate to severe MR. The aim of the current study is to evaluate the Cardioband annuloplasty system for repair the Tricuspid Regurgitation.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic functional tricuspid regurgitation (FTR) with annular diameter ≥ 40 mm with valve Systolic pulmonary pressure (sPAP) ≤ 60mmHg
2. ≥18 years old
3. New York Heart Association (NYHA) Class II-IVa
4. Symptomatic despite Guideline Directed Medical Therapy (GDMT); at minimum patient on diuretic regimen
5. LVEF ≥ 30%
6. Patient is willing and able to comply with all specified study evaluations
7. The Local Site Heart Team concur that surgery will not be offered as a treatment option
8. Transfemoral access of the Cardioband is determined to be feasible

Exclusion Criteria:

1. Aortic, mitral and/or pulmonic valve stenosis and/or regurgitation ≥ moderate
2. Severe uncontrolled hypertension (Systolic BP ≥ 180 mmHg and/or Diastolic BP ≥ 110 mm Hg)
3. Previous tricuspid valve repair or replacement
4. Trans-tricuspid pacemaker or defibrillator leads suggesting impingement of the of the tricuspid valve leaflets, as evaluated by echocardiography
5. Active endocarditis
6. MI or known unstable angina within the 30 days prior to the index procedure
7. Any percutaneous coronary intervention (PCI) or transcatheter valvular intervention within 30 days prior to the index
8. Hemodynamic instability or on IV inotropes
9. Cerebrovascular Accident (CVA) within the past 6 months
10. Subject is on chronic dialysis
11. Anemia (Hb < 9 g/dL) not corrected by transfusion
12. Bleeding disorders or hypercoaguable state
13. Active peptic ulcer or active gastrointestinal (GI) bleeding
14. Contraindication to anticoagulants
15. Known allergy to stainless steel, nickel, and/or polyester
16. Pregnant or lactating; or female of childbearing potential with a positive pregnancy test 24 hours before any study-related radiation exposure
17. In the judgment of the Investigator, co-morbid condition(s) that could limit the subject's ability to participate in the study, including compliance with follow-up requirements, or that could impact the scientific integrity of the study
18. Life expectancy of less than 12 months
19. Impaired judgment and/or is undergoing emergency treatment
20. Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study
21. intra-cardiac masses, thrombi or vegetations
22. Patients with cardiac cachexia
23. Subjects in whom transesophageal echocardiography is contraindicated
24. . Known hypersensitivity or contraindication to procedural medications which cannot be adequately managed medically
25. Untreated clinically significant CAD requiring revascularization
26. Echocardiographic evidence of severe right ventricular dysfunction
27. Any coronary or endovascular surgery, within 3 months prior to procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2018-01-01 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nickenig, MD, Principal Investigator — University Hospital, Bonn
Locations (8):
- Hôpital Bichat-Claude Bernard, Paris, France
- Germany (6):
  - Bonn University - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Köln, Cologne
  - Asklepios Klinik, St. Georg, Hamburg
  - Universitätsklinik Hamburg Eppendorf, Herzzentrum, Hamburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - LMU Klinikum der Universität München, Medizinische Klinik I, Munich
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nickenig G, Weber M, Schuler R, Hausleiter J, Nabauer M, von Bardeleben RS, Sotiriou E, Schafer U, Deuschl F, Alessandrini H, Kreidel F, Juliard JM, Brochet E, Latib A, Montorfano M, Agricola E, Baldus S, Friedrichs KP, Deo SH, Gilmore SY, Feldman T, Hahn RT, Maisano F. Tricuspid valve repair with the Cardioband system: two-year outcomes of the multicentre, prospective TRI-REPAIR study. EuroIntervention. 2021 Feb 5;16(15):e1264-e1271. doi: 10.4244/EIJ-D-20-01107. PMID 33046437
- [Derived] Nickenig G, Weber M, Schueler R, Hausleiter J, Nabauer M, von Bardeleben RS, Sotiriou E, Schafer U, Deuschl F, Kuck KH, Kreidel F, Juliard JM, Brochet E, Latib A, Agricola E, Baldus S, Friedrichs K, Vandrangi P, Verta P, Hahn RT, Maisano F. 6-Month Outcomes of Tricuspid Valve Reconstruction for Patients With Severe Tricuspid Regurgitation. J Am Coll Cardiol. 2019 Apr 23;73(15):1905-1915. doi: 10.1016/j.jacc.2019.01.062. PMID 30999993

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardioband Tricuspid Procedure
Started | 40
Completed | 29
Not Completed | 11
Not completed — Death | 9
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawal to non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Calculated BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.0 (3.9)
STS Score [Mean (Standard Deviation); unit: Percentage of expected mortality] — The STS score is a validated risk-prediction model for open surgery based on data from the STS National Adult Cardiac Surgery Database. In general, an STS predicted risk of surgical mortality of 4%-8% is considered intermediate risk and 8% or greater is considered high risk.
  As of November 15, 2018, The Society of Thoracic Surgeons released an updated short-term risk calculator to reflect the latest 2018 adult cardiac surgery risk models. The STS Calculator allows you to calculate a patient's risk of mortality and morbidities for the most commonly performed cardiac surgeries.
  Percentage of expected mortality | 2.8 (1.5)
EUROSCORE II [Mean (Standard Deviation); unit: Score] — EuroScore II is a risk model which allows the calculation of the risk of death after a heart operation.
  EuroScore II risk levels are as follows:
  * < 8: Low risk
  * 8-10: Moderate risk •>10: High risk
  Score | 4.4 (2.9)
NYHA Class [Count of Participants; unit: Participants] — NYHA Classification - The stages of heart failure:
  1. Class I - No symptoms and no limitation in ordinary physical activity
  2. Class II - Mild symptoms and slight limitation during ordinary activity.
  3. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  4. Class IV - Severe limitations. Experiences symptoms even while at rest.
  Participants
    II | 6
    III | 32
    IV | 2
NYHA Class Grouped [Count of Participants; unit: Participants] — Measure Description: NYHA Classification - The stages of heart failure:
  1. Class I - No symptoms and no limitation in ordinary physical activity
  2. Class II - Mild symptoms and slight limitation during ordinary activity.
  3. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  4. Class IV - Severe limitations. Experiences symptoms even while at rest.
  Participants
    I/II | 6
    III/IV | 34
Left Ventricle Ejection Franction (LVEF) % [Mean (Standard Deviation); unit: Percent Fraction] — Population: The outcome is reported for subjects where data is available. Subjects with missing data are excluded from the analysis.
  Percent Fraction
    number analyzed (Participants) | 38
    (all) | 56.9 (10.2)
FTR Etiology [Count of Participants; unit: Participants]
  Ischemic | 7
  Non-ischemic | 33
Valve Surgery [Count of Participants; unit: Participants]
  Mitral Valve | 4
  Aortic Valve | 1
  Mitral and Aortic Valve | 1
  Other | 0
Percutaneous Transcatheter Valve Replace/Repair other than Tricuspid [Count of Participants; unit: Participants]
  Transcatheter Aortic Valve Implantation | 0
  Mitraclip | 4
  Other | 0
CABG [Count of Participants; unit: Participants]
  Single | 3
  Double | 3
  Triple/Quadruple/Quintuple | 2
Percutaneous Coronary Intervention [Count of Participants; unit: Participants] | 8
Any Cardiac Device without Electrodes [Count of Participants; unit: Participants]
  Parachute Implant | 0
  LAA Closure | 2
  PFO Closure | 1
Any Cardiac Device with Electrodes [Count of Participants; unit: Participants]
  Single Chamber Pacemaker Implant | 1
  Dual Chamber Pacemaker Implant | 3
  CRT Implant | 0
  ICD Implant | 2
  CRT-D Implant | 1
Coronary Artery Disease [Count of Participants; unit: Participants] | 17
Previous MI [Count of Participants; unit: Participants] | 2
Angina Pectoris [Count of Participants; unit: Participants] | 0
Congestive Heart Failure [Count of Participants; unit: Participants] | 25
Aortic Valve [Count of Participants; unit: Participants]
  Moderate Regurgitation | 0
  Severe Regurgitation | 0
  Moderate Stenosis | 0
  Severe Stenosis | 0
  None | 40
Mitral Valve [Count of Participants; unit: Participants]
  Moderate Regurgitation | 0
  Severe Regurgitation | 0
  Moderate Stenosis | 0
  Severe Stenosis | 0
  None | 40
Pulmonic Valve [Count of Participants; unit: Participants]
  Moderate Regurgitation | 0
  Severe Regurgitation | 0
  Moderate Stenosis | 0
  Severe Stenosis | 0
  None | 40
Atrial Flutter/Fibrillation [Count of Participants; unit: Participants]
  None | 3
  Paroxysmal | 5
  Persistant | 20
  Chronic | 12
Flutter/Fibrillation Ablation [Count of Participants; unit: Participants] | 8
Ventricular Tachyarrhthmia [Count of Participants; unit: Participants]
  None | 38
  Sustained | 1
  Non-sustained | 0
  VF | 1
Diabetes [Count of Participants; unit: Participants] | 10
Dyslipidemia [Count of Participants; unit: Participants] | 22
Systemic Hypertension [Count of Participants; unit: Participants] | 33
Peripheral Vascular Disease [Count of Participants; unit: Participants] | 7
Peripheral Vascular Intervention [Count of Participants; unit: Participants] | 0
Chronic Lung Disease (Moderate to Severe) [Count of Participants; unit: Participants] | 11
Chronic Renal Disease [Count of Participants; unit: Participants] | 22
Chronic Liver Disease [Count of Participants; unit: Participants]
  None/Mild | 40
  Moderate | 0
  Severe | 0
Chronic Anemia [Count of Participants; unit: Participants] | 5
Estimated Glomerular Filtration (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 46.3 (17.6)
History of Endocarditis [Count of Participants; unit: Participants] | 1
Thyreosis [Count of Participants; unit: Participants]
  Hyperthyreosis | 0
  Hypothyreosis | 12
Ongoing Inotropic Support [Count of Participants; unit: Participants] | 0
Elevated Pulmonary Pressure (> 35mmHG) [Count of Participants; unit: Participants] | 19
Pulmonary Pressure [Mean (Standard Deviation); unit: mmHg] — Population: The outcome is reported for subjects where data is available. Subjects with missing data are excluded from the analysis.
  mmHg
    number analyzed (Participants) | 37
    (all) | 36.5 (11.5)
Frailty Score [Count of Participants; unit: Participants]
  Very Fit (1) | 0
  Well (2)/Well with Treated Comorbid Disease (3) | 14
  Apparently Vulnerable (4) | 6
  Mildly Frail (5)/Moderately Frail (6) | 20
  Severely Frail (7) | 0
Prior Stroke [Count of Participants; unit: Participants] | 4
Prior Transient Ischemic Attack [Count of Participants; unit: Participants] | 2
Carotid Surgery [Count of Participants; unit: Participants] | 1
Carotid Intervention [Count of Participants; unit: Participants] | 0
History of Smoking [Count of Participants; unit: Participants]
  None | 26
  Current | 3
  Past | 11
Active Malignancy [Count of Participants; unit: Participants] | 0
Other Relevant Medical Conditions [Count of Participants; unit: Participants] | 32

OUTCOME MEASURES:

1. Primary Outcome: Major Serious Adverse Events (MSAEs) and Serious Adverse Device Effects (SADE)
Description: Overall rate of Major Serious Adverse Events (MSAEs)* and serious adverse device effects (SADE)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
Participants
  MSAE | 3
  SADE | 1

2. Primary Outcome: Access, Deployment and Positioning of the Cardioband Device
Description: Successful access, deployment and positioning of the Cardioband device
Time Frame: Intra-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
Participants | 39

3. Secondary Outcome: Technical Success
Description: Successful access, deployment and positioning of the Cardioband device and septolateral reduction.
Time Frame: 1, 6, 12, and 24 months
Population: Data was not collected
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 0

4. Secondary Outcome: Tricuspid Regurgitation [Paired Baseline and Follow-Up]
Description: Data available at each time point was reported as number of patients with TR grades between Trace, Mild, Moderate, and Severe. Data analysis per core lab.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The data is presented as paired data for patients that have baseline data and data for each individual follow up time point. The number of patients with paired data between baseline, 1 month, 30 days, 6 months, 12 months, and 24 months is 37, 33, 37, and 20 respectively. The outcome is reported where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 37
Participants
  Baseline (1 Month): None | 0
  Baseline (1 Month): Mild | 0
  Baseline (1 Month): Moderate | 0
  Baseline (1 Month): Severe | 37
  1 Month: None | 0
  1 Month: Mild | 5
  1 Month: Moderate | 11
  1 Month: Severe | 21
  Baseline (6 Months): number analyzed (Participants) | 33
  Baseline (6 Months): None | 0
  Baseline (6 Months): Mild | 0
  Baseline (6 Months): Moderate | 0
  Baseline (6 Months): Severe | 33
  6 Months: number analyzed (Participants) | 33
  6 Months: None | 0
  6 Months: Mild | 3
  6 Months: Moderate | 10
  6 Months: Severe | 20
  Baseline (12 Months): number analyzed (Participants) | 27
  Baseline (12 Months): None | 0
  Baseline (12 Months): Mild | 0
  Baseline (12 Months): Moderate | 0
  Baseline (12 Months): Severe | 27
  12 Months: number analyzed (Participants) | 27
  12 Months: None | 0
  12 Months: Mild | 2
  12 Months: Moderate | 9
  12 Months: Severe | 16
  Baseline (24 Months): number analyzed (Participants) | 20
  Baseline (24 Months): None | 0
  Baseline (24 Months): Mild | 0
  Baseline (24 Months): Moderate | 0
  Baseline (24 Months): Severe | 20
  24 Months: number analyzed (Participants) | 20
  24 Months: None | 0
  24 Months: Mild | 8
  24 Months: Moderate | 7
  24 Months: Severe | 5

5. Secondary Outcome: Tricuspid Regurgitation [Full Analysis Data Set]
Description: All data available at each time point was reported as number of patients with TR grades between Trace, Mild, Moderate, Severe. Data analysis per core lab.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
Participants
  Baseline: None | 0
  Baseline: Mild | 0
  Baseline: Moderate | 0
  Baseline: Severe | 40
  1 Month: number analyzed (Participants) | 37
  1 Month: None | 0
  1 Month: Mild | 5
  1 Month: Moderate | 11
  1 Month: Severe | 21
  6 Months: number analyzed (Participants) | 33
  6 Months: None | 0
  6 Months: Mild | 3
  6 Months: Moderate | 10
  6 Months: Severe | 20
  12 Months: number analyzed (Participants) | 27
  12 Months: None | 0
  12 Months: Mild | 2
  12 Months: Moderate | 9
  12 Months: Severe | 16
  24 Months: number analyzed (Participants) | 20
  24 Months: None | 0
  24 Months: Mild | 8
  24 Months: Moderate | 7
  24 Months: Severe | 5

6. Secondary Outcome: Effective Regurgitant Orifice Area (EROA) [Paired Baseline and Follow-Up]
Description: Effective regurgitant orifice area (EROA) at 1 month, 6 months, 12 months, and 24 months over baseline. Data analysis per core lab
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The data is presented as paired data for patients that have baseline data and data for each individual follow up time point. The number of patients with paired data between baseline and 1 month, 6 months, 12 months, and 24 months is 28, 21, 18, and 12 respectively. The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 38
cm^2
  Baseline (1 Month): number analyzed (Participants) | 28
  Baseline (1 Month) | 0.8 (0.5)
  1 Month: number analyzed (Participants) | 28
  1 Month | 0.6 (0.6)
  Baseline (6 Months): number analyzed (Participants) | 21
  Baseline (6 Months) | 0.8 (0.5)
  6 Months: number analyzed (Participants) | 21
  6 Months | 0.4 (0.3)
  Baseline (12 Months): number analyzed (Participants) | 18
  Baseline (12 Months) | 0.8 (0.5)
  12 Months: number analyzed (Participants) | 18
  12 Months | 0.4 (0.2)
  Baseline (24 Months): number analyzed (Participants) | 12
  Baseline (24 Months) | 0.3 (0.2)
  24 Months: number analyzed (Participants) | 12
  24 Months | -0.6 (0.4)

7. Secondary Outcome: Effective Regurgitant Orifice Area (EROA) [Full Analysis Data Set]
Description: All data available for Effective regurgitant orifice area (EROA) at 1 month, 6 months, 12 months, and 24 months over baseline. Data analysis per core lab.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
cm^2
  Baseline: number analyzed (Participants) | 34
  Baseline | 0.8 (0.5)
  1 Month: number analyzed (Participants) | 33
  1 Month | 0.6 (0.6)
  6 Months: number analyzed (Participants) | 24
  6 Months | 0.4 (0.3)
  12 Months: number analyzed (Participants) | 19
  12 Months | 0.4 (0.2)
  24 Months: number analyzed (Participants) | 14
  24 Months | 0.3 (0.2)

8. Secondary Outcome: Regurgitant Volume [Paired Baseline and Follow-Up]
Description: Regurgitant Volume (by Echocardiography) data available at 1 month, 6 months, 12 months, and 24 months over baseline. Data analysis per core lab.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The data is presented as paired data for patients that have baseline data and data for each individual follow up time point. The number of patients with paired data between baseline and 1 month, 6 months, 12 months, and 24 months is 11, 12, 3, and 4 respectively.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 38
ml
  Baseline (1 Month): number analyzed (Participants) | 11
  Baseline (1 Month) | 97.1 (35.6)
  1 Month: number analyzed (Participants) | 11
  1 Month | 70.7 (50.5)
  Baseline (6 Months): number analyzed (Participants) | 12
  Baseline (6 Months) | 104.2 (33.5)
  6 Months: number analyzed (Participants) | 12
  6 Months | 76.9 (51.5)
  Baseline (12 Months): number analyzed (Participants) | 3
  Baseline (12 Months) | 76.5 (32.2)
  12 Months: number analyzed (Participants) | 3
  12 Months | 51.2 (16.9)
  Baseline (24 Months): number analyzed (Participants) | 4
  Baseline (24 Months) | 98.1 (41.5)
  24 Months: number analyzed (Participants) | 4
  24 Months | 47.2 (35.3)

9. Secondary Outcome: Regurgitant Volume [Full Analysis Data Set]
Description: All data for Regurgitant Volume (by Echocardiography) at 1 month, 6 months, 12 months, and 24 months over baseline. Data analysis per core lab.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
ml
  Baseline: number analyzed (Participants) | 20
  Baseline | 104.4 (37.0)
  1 Month: number analyzed (Participants) | 20
  1 Month | 86.7 (51.7)
  6 Months: number analyzed (Participants) | 20
  6 Months | 78.4 (43.2)
  12 Months: number analyzed (Participants) | 14
  12 Months | 79.4 (35.4)
  24 Months: number analyzed (Participants) | 5
  24 Months | 56.7 (37.3)

10. Secondary Outcome: TAPSE [Paired Baseline and Follow-Up]
Description: Tricuspid Annular Plane Systolic Excursion at 1 month, 6 months, 12 months, and 24 months over baseline. Data analysis per core lab.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The data is presented as paired data for patients that have baseline data and data for each individual follow up time point. The number of patients with paired data between baseline, 1 month, 6 months, 12 months, and 24 months is 28, 26, 24, and 17 respectively.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 38
cm
  Baseline (30 Days): number analyzed (Participants) | 28
  Baseline (30 Days) | 1.4 (0.4)
  30 Days: number analyzed (Participants) | 28
  30 Days | 1.3 (0.4)
  Baseline (6 Months): number analyzed (Participants) | 26
  Baseline (6 Months) | 1.4 (0.4)
  6 Months: number analyzed (Participants) | 26
  6 Months | 1.4 (0.3)
  Baseline (12 Months): number analyzed (Participants) | 24
  Baseline (12 Months) | 1.4 (0.3)
  12 Months: number analyzed (Participants) | 24
  12 Months | 1.3 (0.3)
  Baseline (24 Months): number analyzed (Participants) | 17
  Baseline (24 Months) | 1.4 (0.4)
  24 Months: number analyzed (Participants) | 17
  24 Months | 1.3 (0.4)

11. Secondary Outcome: TAPSE [Full Analysis Data Set]
Description: All data for Tricuspid Annular Plane Systolic Excursion at 1 month, 6 months, 12 months, and 24 months over baseline. Data analyses based on core lab assessment.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
cm
  Baseline: number analyzed (Participants) | 32
  Baseline | 1.5 (0.3)
  30 Days: number analyzed (Participants) | 35
  30 Days | 1.4 (0.4)
  6 Months: number analyzed (Participants) | 32
  6 Months | 1.4 (0.4)
  12 Months: number analyzed (Participants) | 28
  12 Months | 1.3 (0.3)
  24 Months: number analyzed (Participants) | 21
  24 Months | 1.4 (0.4)

12. Secondary Outcome: NYHA [Paired Baseline and Follow-Up]
Description: NYHA classification data available at 1 month, 6 months, 12 months, 24 months over baseline.
  Measure Description: NYHA Classification - The stages of heart failure:
  1. Class I - No symptoms and no limitation in ordinary physical activity
  2. Class II - Mild symptoms and slight limitation during ordinary activity.
  3. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  4. Class IV - Severe limitations. Experiences symptoms even while at rest.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The data is presented as paired data for patients that have baseline data and data for each individual follow up time point. The number of patients with paired data between baseline, 1 month, 6 months, 12 months, and 24 months is 37, 35, 30, and 25 respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 37
Participants
  Baseline (1 Month): I | 0
  Baseline (1 Month): II | 6
  Baseline (1 Month): III | 30
  Baseline (1 Month): IV | 1
  1 Month: I | 5
  1 Month: II | 22
  1 Month: III | 10
  1 Month: IV | 0
  Baseline (6 Months): number analyzed (Participants) | 35
  Baseline (6 Months): I | 0
  Baseline (6 Months): II | 6
  Baseline (6 Months): III | 28
  Baseline (6 Months): IV | 1
  6 Months: number analyzed (Participants) | 35
  6 Months: I | 8
  6 Months: II | 19
  6 Months: III | 8
  6 Months: IV | 0
  Baseline (12 Months): number analyzed (Participants) | 30
  Baseline (12 Months): I | 0
  Baseline (12 Months): II | 6
  Baseline (12 Months): III | 23
  Baseline (12 Months): IV | 1
  12 Months: number analyzed (Participants) | 30
  12 Months: I | 10
  12 Months: II | 12
  12 Months: III | 7
  12 Months: IV | 1
  Baseline (24 Months): number analyzed (Participants) | 25
  Baseline (24 Months): I | 0
  Baseline (24 Months): II | 5
  Baseline (24 Months): III | 20
  Baseline (24 Months): IV | 0
  24 Months: number analyzed (Participants) | 25
  24 Months: I | 6
  24 Months: II | 12
  24 Months: III | 7
  24 Months: IV | 0

13. Secondary Outcome: NYHA [Full Analysis Data Set]
Description: All data available for NYHA classification at 1 month, 6 months, 12 months, and 24 months over baseline.
  Measure Description: NYHA Classification - The stages of heart failure:
  1. Class I - No symptoms and no limitation in ordinary physical activity
  2. Class II - Mild symptoms and slight limitation during ordinary activity.
  3. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  4. Class IV - Severe limitations. Experiences symptoms even while at rest.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
Participants
  Baseline: I | 0
  Baseline: II | 6
  Baseline: III | 32
  Baseline: IV | 2
  1 Month: number analyzed (Participants) | 37
  1 Month: I | 5
  1 Month: II | 22
  1 Month: III | 10
  1 Month: IV | 0
  6 Months: number analyzed (Participants) | 35
  6 Months: I | 8
  6 Months: II | 19
  6 Months: III | 8
  6 Months: IV | 0
  12 Months: number analyzed (Participants) | 30
  12 Months: I | 10
  12 Months: II | 12
  12 Months: III | 7
  12 Months: IV | 1
  24 Months: number analyzed (Participants) | 25
  24 Months: I | 6
  24 Months: II | 12
  24 Months: III | 7
  24 Months: IV | 0

14. Secondary Outcome: 6MWT [Paired Baseline and Follow-Up]
Description: Distance in meters walked during 6 Minute Walk Test (6MWT) at 1 month, 6 months, 12 months, and 24 months over baseline.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The data is presented as paired data for patients that have baseline data and data for each individual follow up time point. The number of patients with paired data between baseline and 1 month, 6 months, 12 months, and 24 months is 29, 28, 25, and 17 respectively.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 29
Meters
  Baseline (1 Month) | 232.0 (117.5)
  1 Month | 289.4 (118.7)
  Baseline (6 Months): number analyzed (Participants) | 28
  Baseline (6 Months) | 236.1 (107.8)
  6 Months: number analyzed (Participants) | 28
  6 Months | 280.6 (132.8)
  Baseline (12 Months): number analyzed (Participants) | 25
  Baseline (12 Months) | 222.2 (104.7)
  12 Months: number analyzed (Participants) | 25
  12 Months | 273.6 (133.4)
  Baseline (24 Months): number analyzed (Participants) | 17
  Baseline (24 Months) | 211.6 (124.9)
  24 Months: number analyzed (Participants) | 17
  24 Months | 294.3 (121.0)

15. Secondary Outcome: 6MWT [Full Analysis Data Set]
Description: Distance in meters walked during 6 minute walk test (6MWT) at 1 month, 6 months, 12 months, and 24 months over baseline.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 36
Meters
  Baseline | 221.9 (113.0)
  1 Month: number analyzed (Participants) | 29
  1 Month | 289.4 (118.7)
  6 Months: number analyzed (Participants) | 29
  6 Months | 279.2 (130.6)
  12 Months: number analyzed (Participants) | 25
  12 Months | 273.6 (133.4)
  24 Months: number analyzed (Participants) | 18
  24 Months | 288.2 (120.2)

16. Secondary Outcome: Kansas City Cardiomyopathy (KCCQ) [Paired Baseline and Follow-Up]
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ-12) is a self-administered, 12-item questionnaire that quantifies physical limitations, symptoms, self-sufficiency, social interaction and quality of life. Scores range from 0-100, in which higher scores reflect better health status. An increase in the KCCQ-12 score reflects an improvement in symptoms for the subject. A mean difference over time of 5 points on the KCCQ-12 summary score reflects a clinically significant change in heart failure status.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The data is presented as paired data for patients that have baseline data and data for each individual follow up time point. The number of patients with paired data between baseline and 1 month, 6 months, 12 months, and 24 months is 37, 35, 31, and 28 respectively.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 37
Score
  Baseline (1 Month) | 44.4 (21.8)
  1 Month | 56.7 (24.0)
  Baseline (6 Months): number analyzed (Participants) | 35
  Baseline (6 Months) | 44.6 (21.1)
  6 Months: number analyzed (Participants) | 35
  6 Months | 63.6 (23.8)
  Baseline (12 Months): number analyzed (Participants) | 31
  Baseline (12 Months) | 43.3 (21.6)
  12 Months: number analyzed (Participants) | 31
  12 Months | 59.6 (22.7)
  Baseline (24 Months): number analyzed (Participants) | 28
  Baseline (24 Months) | 47.0 (20.9)
  24 Months: number analyzed (Participants) | 28
  24 Months | 58.0 (24.3)

17. Secondary Outcome: Kansas City Cardiomyopathy (KCCQ) [Full Analysis Data Set]
Description: as for outcome 16
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
units on a scale
  Baseline | 43.8 (21.9)
  1 Month: number analyzed (Participants) | 37
  1 Month | 56.7 (24.0)
  6 Months: number analyzed (Participants) | 35
  6 Months | 63.6 (23.8)
  12 Months: number analyzed (Participants) | 31
  12 Months | 59.6 (22.7)
  24 Months: number analyzed (Participants) | 28
  24 Months | 58.0 (24.3)

18. Secondary Outcome: Left Ventricle Ejection Fraction (LVEF) [Paired Baseline and Follow-Up]
Description: Left ventricle ejection fraction data available for 1 month, 6 months, 12 months, and 24 months over baseline. Data analysis based on core lab assessment.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The data is presented as paired data for patients that have baseline data and data for each individual follow up time point. The number of patients with paired data between baseline and 1 month, 6 months, 12 months, and 24 months is 31, 30, 25, and 19 respectively.
Measure: Mean (Standard Deviation); unit: percent fraction
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 38
percent fraction
  Baseline (1 Month): number analyzed (Participants) | 31
  Baseline (1 Month) | 56.7 (10.0)
  1 Month: number analyzed (Participants) | 31
  1 Month | 57.0 (8.4)
  Baseline (6 Months): number analyzed (Participants) | 30
  Baseline (6 Months) | 56.2 (10.0)
  6 Months: number analyzed (Participants) | 30
  6 Months | 57.4 (7.1)
  Baseline (12 Months): number analyzed (Participants) | 25
  Baseline (12 Months) | 56.6 (10.1)
  12 Months: number analyzed (Participants) | 25
  12 Months | 58.8 (6.5)
  Baseline (24 Months): number analyzed (Participants) | 19
  Baseline (24 Months) | 57.8 (8.8)
  24 Months: number analyzed (Participants) | 19
  24 Months | 56.6 (6.6)

19. Secondary Outcome: Left Ventricle Ejection Fraction (LVEF) [Full Analysis Data Set]
Description: All available data for left ventricle ejection fraction at 1 month, 6 months, 12 months, and 24 months over baseline. Data analysis per echo core lab.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: percent fraction
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
percent fraction
  Baseline: number analyzed (Participants) | 38
  Baseline | 56.9 (10.2)
  1 Month: number analyzed (Participants) | 32
  1 Month | 57.0 (8.3)
  6 Months: number analyzed (Participants) | 32
  6 Months | 57.8 (7.1)
  12 Months: number analyzed (Participants) | 27
  12 Months | 59.0 (6.3)
  24 Months: number analyzed (Participants) | 20
  24 Months | 56.9 (6.5)

20. Secondary Outcome: Left Ventricle End Diastolic Volume Index (LVEDVI) [Full Analysis Data Set]
Description: Left ventricle end diastolic volume index data available for 1 month, 6 months, 12 months, and 24 months over baseline.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: Data was not collected.
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 0

21. Secondary Outcome: Left Ventricle End Systolic Volume Index (LVESVI) [Full Analysis Data Set]
Description: Left ventricle end systolic volume index data available at 1 month, 6 months, 12 months, and 24 months over baseline.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: Data was not collected.
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 0

22. Secondary Outcome: NT-pro BNP [Full Analysis Data Set]
Description: N-terminal prohormone of brain natriuretic peptide data available at 1 month, 6 months, 12 months, and 24 months over baseline.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
ng/L
  Baseline: number analyzed (Participants) | 32
  Baseline | 2899.3 (2632.5)
  1 Month: number analyzed (Participants) | 28
  1 Month | 2874.5 (2860.5)
  6 Months: number analyzed (Participants) | 30
  6 Months | 2563.1 (2510.2)
  12 Months: number analyzed (Participants) | 24
  12 Months | 2095.5 (2306.4)
  24 Months: number analyzed (Participants) | 18
  24 Months | 2119.1 (2461.3)

23. Secondary Outcome: Diuretic Therapy
Description: Diuretic Therapy data available at 1 month, 6 months, 12 months, and 24 months over baseline.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: Data was not collected.
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 0

24. Secondary Outcome: Bilirubin [Full Analysis Data Set]
Description: Bilirubin data available at 1 month, 6 months, 12 months, and 24 months over baseline.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
umol/L
  Bilirubin Baseline: number analyzed (Participants) | 36
  Bilirubin Baseline | 15.7 (17.5)
  Bilirubin 1 Month: number analyzed (Participants) | 32
  Bilirubin 1 Month | 14.0 (13.4)
  Bilirubin 6 Months: number analyzed (Participants) | 36
  Bilirubin 6 Months | 13.0 (5.8)
  Bilirubin 12 Months: number analyzed (Participants) | 27
  Bilirubin 12 Months | 11.6 (7.9)
  Bilirubin 24 Months: number analyzed (Participants) | 17
  Bilirubin 24 Months | 7.4 (6.0)

25. Secondary Outcome: Blood Urea Nitrogen (BUN), Serum Creatinine [Full Analysis Data Set]
Description: All available data for Blood urea nitrogen (BUN) and Serum Creatinine at 1 month, 6 months, 12 months, and 24 months over baseline.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
mg/dL
  Baseline: number analyzed (Participants) | 39
  Baseline | 52.8 (30.3)
  1 Month: number analyzed (Participants) | 34
  1 Month | 52.1 (36.0)
  6 Months: number analyzed (Participants) | 36
  6 Months | 64.2 (55.1)
  12 Months: number analyzed (Participants) | 28
  12 Months | 49.5 (34.5)
  24 Months: number analyzed (Participants) | 19
  24 Months | 50.5 (55.7)

26. Secondary Outcome: Activity by Wearable Device
Description: Activity by wearable device available data at 1 month, 6 months, 12 months, and 24 months over baseline.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: Data was not collected.
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 0

27. Secondary Outcome: Glutamic Oxaloacetic Transaminase (GOT) Aspartate Transaminase (AST) [Full Analysis Data Set]
Description: All data available for Glutamic oxaloacetic transaminase (GOT) and Aspartate Transaminase (AST) at 1 month, 6 months, 12 months, and 24 months over baseline.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
U/L
  Baseline: number analyzed (Participants) | 39
  Baseline | 28.3 (9.5)
  1 Month: number analyzed (Participants) | 33
  1 Month | 31.9 (18.3)
  6 Months: number analyzed (Participants) | 36
  6 Months | 30.9 (21.3)
  12 Months: number analyzed (Participants) | 29
  12 Months | 32.3 (10.9)
  24 Months: number analyzed (Participants) | 21
  24 Months | 27.6 (9.6)

28. Secondary Outcome: Glutamic Pyruvic Transaminase (GPT) Alanine Transaminase (ALT) [Full Analysis Data Set]
Description: All data available for glutamic pyruvic transaminase (GPT) Alanine Transaminase (ALT) at 1 month, 6 months, 12 months, and 24 months.
Time Frame: 1, 6, 12, and 24 months over baseline
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Cardioband Tricuspid Procedure
Number analyzed (Participants) | 40
IU/L
  Baseline | 21.9 (14.0)
  1 Month: number analyzed (Participants) | 34
  1 Month | 25.1 (23.8)
  6 Months: number analyzed (Participants) | 36
  6 Months | 23.4 (18.4)
  12 Months: number analyzed (Participants) | 29
  12 Months | 24.6 (12.2)
  24 Months: number analyzed (Participants) | 24
  24 Months | 18.6 (10.2)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cardioband Tricuspid Procedure
All-Cause Mortality (participants affected / at risk) | 9/40
Serious Adverse Events (participants affected / at risk) | 33/40
Other Adverse Events (participants affected / at risk) | 34/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardioband Tricuspid Procedure (N=40)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Chronic lymphocytic leukaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 13 (19)
Tricuspid valve incompetence (Cardiac disorders) | 6 (6)
Atrioventricular block complete (Cardiac disorders) | 3 (3)
Right ventricular failure (Cardiac disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Chronotropic incompetence (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Coronary artery perforation (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Diabetic foot infection (Endocrine disorders) | 1 (1)
Hyperglycaemia (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Diverticulosis (Gastrointestinal disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Jejunal ulcer (Gastrointestinal disorders) | 1 (1)
MalloryWeiss Syndrome (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Erysipelothrix infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Femur Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1)
Somatic symptom disorder (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Cardiopulmonary failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 2 (2)
Syncope (Vascular disorders) | 1 (4)
Haematoma (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
Stasis dermatitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardioband Tricuspid Procedure (N=40)
Anaemia (Blood and lymphatic system disorders) | 9 (10)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (4)
Arteriospasm coronary (Cardiac disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 5 (6)
Atrioventricular block complete (Cardiac disorders) | 3 (3)
Cardiac failure (Cardiac disorders) | 13 (20)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 3 (3)
Right ventricular failure (Cardiac disorders) | 4 (5)
Tricuspid valve incompetence (Cardiac disorders) | 8 (8)
Ventricular tachycardia (Cardiac disorders) | 3 (4)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 2 (2)
Melaena (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Impaired healing (General disorders) | 2 (2)
Infection (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 8 (11)
Fall (Injury, poisoning and procedural complications) | 2 (5)
Postoperative delirium (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Blood thyroid stimulating hormone decreased (Investigations) | 3 (3)
Brain natriuretic peptide increased (Investigations) | 2 (2)
C-reactive protein increased (Investigations) | 3 (3)
Haemoglobin decreased (Investigations) | 5 (5)
Troponin increased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Cerebrovascular accident (Nervous system disorders) | 2 (3)
Device dislocation (Product Issues) | 4 (4)
Device malfunction (Product Issues) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 12 (16)
Chronic Kidney disease (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Haematoma (Vascular disorders) | 2 (3)
Haemorrhage (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT02981953/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT02981953/SAP_001.pdf